CLINICAL TRIAL: NCT01558024
Title: The Effects of Compression Stockings on Pressure Parameters in Patients With Chronic Venous Insufficiency
Acronym: MACIVC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: AOI/2011/APM-03; 2014-A00737-40 (Other: ANSM)
Record Dates: First submitted 2012-03-16; First posted 2012-03-20 (Estimated); Last update posted 2025-12-22 (Actual); Status verified 2016-05

CONDITIONS: Venous Insufficiency
Keywords: compression stockings; physiopathology
MeSH Terms: conditions — Venous Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- C1S patients (Experimental): 18 Patients with venous insufficiency: "C1S" patients according to the CEAP (Clinical-Etiology-Anatomy-Pathophysiology)classification.
  Interventions: Other: Intravenous pressure and intramuscular pressure measurement
- C3 patients (Experimental): 18 Patients with venous insufficiency: "C3" patients according to the CEAP (Clinical-Etiology-Anatomy-Pathophysiology)classification.
  Interventions: Other: Intravenous pressure and intramuscular pressure measurement
- C5 patients (Experimental): 18 Patients with venous insufficiency: "C5" patients according to the CEAP (Clinical-Etiology-Anatomy-Pathophysiology)classification.
  Interventions: Other: Intravenous pressure and intramuscular pressure measurement
- Sedentary volunteers (Experimental): 18 healthy volunteers with a sedentary lifestyle (< 2h of physical activity per week)
  Interventions: Other: Intravenous pressure and intramuscular pressure measurement
- Active volunteers (Experimental): 18 healthy volunteers with an active lifestyle (between 2 and 6 hours of physical activity per week)
  Interventions: Other: Intravenous pressure and intramuscular pressure measurement
- Athletic volunteers (Experimental): 18 healthy volunteers with an athletic lifestyle (over 6 hours of physical activity per week for at least one year)
  Interventions: Other: Intravenous pressure and intramuscular pressure measurement

INTERVENTIONS:
Other: Intravenous pressure and intramuscular pressure measurement — Ultrasound using the Logiq-e system (GE Ultrasound, Chicago, Ill), with a 12L-RS linear probe equipped with a XFTC300 sensor connected to an ARD154 amplifier

SUMMARY:
The main objective of this study is to obtain data to determine, in each individual with and without wearing compression stockings of different strengths and during different postures, the relationship between interface pressure and the area and circumference of the great saphenous vein and posterior tibial veins in the calf and ankle.

ELIGIBILITY:
Inclusion Criteria:

* The participant must have given his/her informed and signed consent
* The participant must be insured or beneficiary of a health insurance plan

Inclusion criteria for patients in the venous insufficiency group:

* CEAP (Clinical-Etiology-Anatomy-Pathophysiology) Classification : C1S, C3 or C5

Inclusion criteria for healthy volunteers

* general good health
* subgroups including:
* sedentary volunteers (< 2hours of physical activity per week)
* active volunteers (between 2 and 6 hours of physical activity per week)
* athletic volunteers (over 6 hours of physical activity per week for at least 1 year)

Exclusion Criteria:

* The participant is participating in another study, except the "volumetric" counterpart to the present study
* The participant is in an exclusion period determined by a previous study
* The participant is under judicial protection, under tutorship or curatorship
* The participant refuses to sign the consent
* It is impossible to correctly inform the participant
* The participant is pregnant, parturient, or breastfeeding
* Arterial vascular disease, heart, lymph, renal, hepatic, oncologic, metabolic or endocrine or any other condition that may cause or exaggerate edema

Exclusion criteria for healthy volunteers:

* Risk for abnormal bleeding (hemophilia, anticoagulation or antiplatelet)
* Taking diuretics or corticoids

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2014-07; Primary Completion 2016-03-31 (Actual); Study Completion 2016-03-31 (Actual)

PRIMARY OUTCOMES:
Correlation between D and A/F at the calf | Baseline (Day 0)
  D = the diameters of the largest cross section of the posterior tibial veins at calf level; A = the area of the largest cross section of the posterior tibial veins at the calf level; F = interface pressure measured along the leg using a 13 captor system.

SECONDARY OUTCOMES:
Interface pressure for the leg | baseline; day 0
  Interface pressure (mmHg) measured using 13 captors over the entire leg in the following positions: decubitus dorsal, sitting, orthostatic and orthodynamic.
Calf interstitial pressure | base line; day 0
  Intramuscular interstitial pressure is measured in the calf for 1/3 or randomly selected participants in the following positions: decubitus dorsal, sitting, orthostatic and orthodynamic.
Venous pressure at the ankle (mmHg) | baseline; day 0
  Pressure of the great saphenous vein is measured at the ankle in the following positions: decubitus dorsal, sitting, orthostatic and orthodynamic
Saphenous vein area, calf | baseline, day 0
  Area (mm^2)of the largest cross section of the great saphenous vein at calf level and for the following positions: decubitus dorsal, sitting, orthostatic
Saphenous vein area, ankle | baseline, day 0
  Area (mm^2)of the largest cross section of the great saphenous vein at ankle level and for the following positions: decubitus dorsal, sitting, orthostatic
Posterior tibial vein area, calf | baseline, day 0
  Area (mm^2)of the largest cross section of the posterior tibial veins at calf level and for the following positions: decubitus dorsal, sitting, orthostatic
Posterior tibial vein area, ankle | baseline, day 0
  Area (mm^2)of the largest cross section of the posterior tibial veins at ankle level and for the following positions: decubitus dorsal, sitting, orthostatic
Saphenous vein perimeter, calf | baseline, day 0
  Perimeter (mm)of the largest cross section of the great saphenous vein at calf level and for the following positions: decubitus dorsal, sitting, orthostatic
Saphenous vein perimeter, ankle | baseline, day 0
  Perimeter (mm)of the largest cross section of the great saphenous vein at ankle level and for the following positions: decubitus dorsal, sitting, orthostatic
Posterior tibial vein perimeter, calf | baseline, day 0
  Perimeter (mm)of the largest cross section of the posterior tibial veins at calf level and for the following positions: decubitus dorsal, sitting, orthostatic
Posterior tibial vein perimeter, ankle | baseline, day 0
  Perimeter (mm)of the largest cross section of the posterior tibial veins at ankle level and for the following positions: decubitus dorsal, sitting, orthostatic
Heart height difference (mm); saphenous vein, calf | baseline, day 0
  The difference in height (mm) between the right atrium and the target cross section on the saphenous vein in the following positions: decubitus dorsal, sitting, orthostatic.
Heart height difference (mm); saphenous vein, ankle | baseline, day 0
  The difference in height (mm) between the right atrium and the target cross section on the saphenous vein in the following positions: decubitus dorsal, sitting, orthostatic.
Heart height difference (mm); posterior tibial veins, calf | baseline, day 0
  The difference in height (mm) between the right atrium and the target cross section on the posterior tibial veins in the following positions: decubitus dorsal, sitting, orthostatic.
Heart height difference (mm); posterior tibial vein, ankle | baseline, day 0
  The difference in height (mm) between the right atrium and the target cross section on the posterior tibial veins in the following positions: decubitus dorsal, sitting, orthostatic.
Leg circumference (mm) | baseline; Day 0
  The circumference of the leg is measured every 5 cm in a decubitus dorsal position.

CONTACTS AND LOCATIONS:
Overall Officials: Antonia Perez Martin, MD PhD, Principal Investigator — Centre Hospitalier Universitaire de Nîmes
Locations (2):
- France (2):
  - CHU de Montpellier - Hôpital Saint-Eloi, Montpellier
  - CHU de Nîmes - Hôpital Universitaire Carémeau, Nîmes

REFERENCES:
- [Result] Mestre S, Triboulet J, Demattei C, Veye F, Nou M, Perez-Martin A, Dauzat M, Quere I. Noninvasive measurement of venous wall deformation induced by changes in transmural pressure shows altered viscoelasticity in patients with chronic venous disease. J Vasc Surg Venous Lymphat Disord. 2021 Jul;9(4):987-997.e2. doi: 10.1016/j.jvsv.2020.11.010. Epub 2020 Nov 21. PMID 33227457
- [Derived] Mestre S, Triboulet J, Demattei C, Veye F, Nou M, Perez-Martin A, Dauzat M, Quere I. Acute effects of graduated and progressive compression stockings on leg vein cross-sectional area and viscoelasticity in patients with chronic venous disease. J Vasc Surg Venous Lymphat Disord. 2022 Jan;10(1):186-195.e25. doi: 10.1016/j.jvsv.2021.03.021. Epub 2021 May 6. PMID 33964512